CLINICAL TRIAL: NCT06132932
Title: A Phase Ib/IIa Study to Evaluate the Safety and Preliminary Efficacy of WX390, a PI3K/mTOR Dual Inhibitor, for the Treatment of Advanced Solid Tumors With PIK3CA Mutations
Brief Title: A Study of WX390 in Patients With Advanced Solid Tumors With PIK3CA Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JYA0102
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: PIK3CA Mutation-Related Tumors

STUDY DESIGN:
Intervention Model Description: WX390 continuous oral dosing (1.1 mg once a day).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX390 (Experimental): Participants will receive WX390 continuous oral dosing (1.1 mg once a day).
  Interventions: Drug: WX390

INTERVENTIONS:
Drug: WX390 — Participants will receive WX390 1.1 mg tablet orally once a day for a continuous 28-day cycle.
  Other Names: WXFL10030390

SUMMARY:
The goal of this clinical trial is to evaluate the safety and preliminary efficacy of WX390 in patients with advanced solid tumors. The main question it aims to answer is:

• safety and preliminary efficacy in WX390 therapy. Participants will be treated with WX390 orally and follow the efficacy and safety evaluation according to the protocol.

DETAILED DESCRIPTION:
This study is a multicenter, open-label phase Ib/IIa clinical trial for patients with advanced solid tumors who have failed standard treatment. The study adopts a basket design, divided into 6 cohorts, with a total of 70-80 advanced solid tumor patients with PIK3CA mutations enrolled. Participants will receive WX390 treatment administered continuously daily, with each cycle lasting 28 days, until disease progression or intolerable toxicity occurs. During the study, safety and efficacy will be evaluated, with efficacy assessment based on RECIST 1.1. In addition, the study will collect tumor tissue or blood samples from the participants to explore the relationship between other biomarkers and treatment efficacy, as well as the impact of changes in PIK3CA mutation status before and after treatment on efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Histologically or cytologically confirmed advanced malignant solid tumors (excluding non-small cell lung cancer) who have failed standard treatment, have no standard treatment options, or for whom standard treatment is not suitable at the current stage (colorectal cancer patients must provide genetic test results confirming KRAS wild-type)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of more than 3 months
* At least one measurable lesion according to RECIST 1.1
* Adequate organic function
* Signed and dated informed consent

Exclusion Criteria:

* Anti-tumor treatments such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, or immunotherapy received within 4 weeks before the first use of the study drug
* Other unapproved clinical trial drugs or treatments received within 4 weeks before the first use of the study drug
* Major organ surgery (excluding biopsy) or significant trauma within 4 weeks before the first use of the study drug
* Systemic use of corticosteroids or other immunosuppressive agents within 14 days before the first use of the study drug
* Previous treatment with PI3K, AKT, or mTOR inhibitors
* Active infection requiring systemic anti-infection treatment
* Known alcohol or drug dependence
* Individuals with mental disorders or poor compliance
* Pregnant or lactating women
* The researcher believes that the subject has other serious systemic medical history or other reasons that make them unsuitable for participating in this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Safety of WX390 in treating patients with advanced malignant solid tumors harboring PIK3CA mutations. | From the start of the trial,up to 24 weeks
  Safety will be evaluated by monitoring AE/SAE
Objective Response Rate (ORR) | From the start of the trial,up to 24 weeks
  ORR is defined as the proportion of patients with complete response (CR) and partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) determined according to RECIST 1.1 criteria | From the start of the trial,up to 24 weeks
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD) according to RECIST 1.1.
Duration of Response (DOR) determined according to RECIST 1.1 criteria | From the start of the trial,up to 24 weeks
  DOR is defined as the time from the initial occurrence of a complete response (CR) or partial response (PR) until disease progression or death due to any cause.
Progression-Free Survival (PFS) determined according to RECIST 1.1 criteria | From the start of the trial,up to 24 weeks
  PFS is defined as the time from randomization until objective tumor progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China